CLINICAL TRIAL: NCT04917510
Title: Evaluating the Efficacy of Erector Spinae Block in Routine Hip Arthroscopy: A Prospective Analysis
Brief Title: Evaluating the Efficacy of Erector Spinae Block in Routine Hip Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-21-1223
Record Dates: First submitted 2021-05-28; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Hip Disease; Postoperative Pain
Keywords: Hip; Pain; Arthroscopy
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either the study group or control group prior to undergoing surgery
Who Masked: Participant
Masking Description: Erector spinae block will be performed after general anesthesia has been induced. Patients will be unaware which arm of the study they are in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Will not receive erector spinae block. Will be administered 30 mL of 0.5% Marcaine w/ epinephrine as a local block at the surgical site at the conclusion of the procedure.
  Interventions: Procedure: Local block
- Study (Experimental): Will receive an erector spinae block prior to surgery using 30-45 mL of 0.25 bupivacaine w/ epinephrine and 5 mL of dexmedetomidine. Will be administered 30 mL of 0.5% marcaine w/ epinephrine as a local block at the surgical site at the conclusion of the procedure.
  Interventions: Procedure: Erector spinae block; Procedure: Local block

INTERVENTIONS:
Procedure: Erector spinae block — See experimental arm group description
  Arms: Study
Procedure: Local block — See control and study arm group descriptions for the local block

SUMMARY:
The aim of this project is to evaluate the efficacy of preoperative erector spinae blocks in arthroscopic hip surgery. This will be a prospective randomized controlled trial.

DETAILED DESCRIPTION:
The aim of this project is to evaluate the efficacy of preoperative erector spinae blocks in arthroscopic hip surgery. This will be a prospective randomized controlled trial. The control group will not receive a preoperative block prior to surgery, but will receive local anesthetic at the surgical site at the conclusion of the surgery. The study group will receive a preoperative block and local anesthetic. The primary outcomes will be pain levels and opioid consumption in the post-operative care unit. The secondary outcomes will be pain levels and opioid consumption post-operatively, and functional outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hip arthroscopy for femoroacetabular impingement
* Ages 13-50
* Individuals who have the capacity to provide consent or assent for themselves

Exclusion Criteria:

* Hip arthroscopy for any other reason (not undergoing labral repair, acetabuloplasty, and femoral osteochondroplasty)
* Revision surgery
* Known narcotic use in the 6 months prior to surgery
* Workman's compensation patient
* Pregnancy

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Post Anesthesia Care Unit Opioids | 6 hours post-operatively
  Total morphine milligram equivalents of administered in the post-operative care unit
Post Anesthesia Care Unit Pain | 6 hours post-operatively
  Visual analogue pain score at the time of discharge from the Post Anesthesia Care Unit in which 0 equals no pain and 10 equals extreme pain

SECONDARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score | 1 year post-operatively
  Hip disability and Osteoarthritis Outcome score at post-op visits in which 0 equals no pain and 100 equals unbearable pain
Patient Reported Outcomes measurement Information System Score | 1 year post-operatively
  Patient Reported Outcomes measurement Information System score at post-op visits in which 0 equals no pain and 10 equals extreme pain
Range Of Motion | 1 year post-operatively
  Hip range of motion in degrees of motion, will be examined by the operative surgeon in the office measured by flexion 0-110 degrees with 0 being no range of motion and 110 being full range of motion, internal rotation -5-25 degrees with -5 being no range of motion and -25 being full range of motion, and external rotation 0-60 degrees with 0 being no range of motion and 60 being full range of motion.
Outpatient Opioids | 4 weeks post discharge
  Opioids consumed after discharge from hospital
Outpatient Visual Analog Scale scores | 4 weeks post discharge
  Pain scores each day for the first 4 weeks after surgery on the Visual Analog Scale in which 0 equals no pain and 10 equals unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Coobs, MD, Principal Investigator — Carilion Clinic Ortho Surgeon
Locations (1):
- Institute for Orthopedics and Neurosciences, Roanoke, Virginia, United States